CLINICAL TRIAL: NCT06374732
Title: Effectiveness of a School-based High-intensity Interval Training Intervention in Adolescents: the PRO-HIIT Cluster Randomised Controlled Trial
Brief Title: The Benefits of a High-intensity Interval Training Intervention Delivered in a School Setting Among Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: China Scholarship Council (Unknown); Ningbo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TY2024002
Record Dates: First submitted 2024-03-20; First posted 2024-04-19 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: school; adolescents; high-intensity interval training; randomised control trial; physical activity
MeSH Terms: conditions — Motor Activity | interventions — High-Intensity Interval Training; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity interval training group (Experimental): The experimental group, which will perform high-intensity interval training (HIIT), 5 time per week for 12 weeks.
  Interventions: Behavioral: High-intensity interval training
- Control group (Active Comparator): Control group, which will continue their normal physical activity, including their usual physical education classes.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: High-intensity interval training — The experimental group will perform 6-to-10-minute of high-intensity interval training at the beginning of their physical education lessons or physical activity lessons.
  Arms: High-intensity interval training group
Behavioral: Control group — The control group will maintain their normal behaviour, including regular physical education lessons and physical activity lessons.
  Arms: Control group

SUMMARY:
A 12-week school-based high-intensity interval training intervention, with 8 classes of year 7 students randomly allocated to either intervention or control group. The interval training sessions will last for 6 to 10 minutes and will be delivered 5 times per week. Outcome variables will be physical activity, body composition, cardiorespiratory fitness, muscular strength, bone health, executive function, mental wellbeing, and academic performance, which will be measured pre- and post-intervention and two months after the intervention has been completed.

DETAILED DESCRIPTION:
The purpose of this study is to: 1) evaluate the effectiveness of a 12-week school-based HIIT intervention on cardiorespiratory fitness (primary outcome), physical activity, body composition, muscular strength, bone health, executive function, wellbeing, enjoyment, affect, self-efficacy and academic performance among 12-13-year-old adolescents; 2) to examine the changes of these outcomes following a two-month unstructured summer holiday after the study has been completed; 3) to conduct a process evaluation for the study.

The study is a 12-week high-intensity interval training intervention, which is 6 to 10-minute in length and will be delivered 5 times per week among year 7 adolescents, at the start of physical education and physical activity lessons. We will examine the effectiveness of this intervention on outcomes, such as body composition, cardiorespiratory fitness, muscular health, bone health, cognitive function, mental wellbeing, and academic performance. In addition, The investigators will evaluate the fitness changes between school days (structured day) and a two-month summer holiday (unstructured days). This will be achieved by collecting data at three timepoints: pre- and post-intervention and after a 2-month (summer holiday) following the completion of the intervention.

The high-intensity interval training includes resistance-based exercises, such as jumping jacks, high knees, burpees, squat jumps, lunge jumps, and mountain climbers.

ELIGIBILITY:
Inclusion Criteria:

• Year 7 students

Exclusion Criteria:

* Unable to perform high-intensity exercises due to existing medical contraindications
* Unable to understand the study procedures and provide consent

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 369 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory fitness | Changes from baseline to immediately after the intervention and two month following the cessation of the intervention.
  Cardiorespiratory fitness will be measured using 20-metre shuttle run. The 20-meter shuttle run requires participants to run back and forth between two lines positioned 20 meters apart. To complete a shuttle, participants must reach the other end before a designated beep sounds. The beep is set to allow the participants to start at 8.5 km/h and increase the speed by 0.5 km/h as indicated by a triple beep. The test concludes if a participant fails to complete two consecutive shuttles or volitionally discontinues.

SECONDARY OUTCOMES:
Muscular strength | Changes from baseline to immediately after the intervention and two month following the cessation of the intervention.
  Upper and lower body strength will be assessed using hand grip and standing long jump, respectively. A digital dynamometer with an adjustable grip, with participants standing and elbow in 90-degree flexion, will be employed for measuring the upper body strength in kilogrammes. The test will be performed twice on both hands and an averaged number of the four measurements will be used for reporting. Standing long jump will be measured with an electrical tester, which has high sensitivity and greatly improved accuracy. Participants stand behind the start line with their feet apart and are allowed to swing their arms quickly to jump as far as possible. Each participant will have three attempts, with the best one recorded.
Wellbeing | Changes from baseline to immediately after the intervention and two month following the cessation of the intervention.
  The Chinese version of Strengths and Difficulties Questionnaire (SDQ) will be used to assess the behavioural and emotional outcomes of participants.
Enjoyment | Changes from baseline to immediately after the intervention and two month following the cessation of the intervention.
  Enjoyment of physical activity will be measured using physical activity enjoyment scale.
Motivation | Changes from baseline to immediately after the intervention and two month following the cessation of the intervention.
  Motivation to autonomously engage in physical activity will be assessed using a modified Behaviour Regulation in Exercise Questionnaire.
Affect | Changes from baseline to immediately after the intervention and two month following the cessation of the intervention.
  Affect will be assessed via a Chinese version of the International Positive and Negative Affect Schedule Short Form
Academic performance | Baseline and immediately after the intervention
  Academic performance will be evaluated by utilising the school's end-of-term academic examinations. The total score for the academic examinations of each participant during term one (January 2023) and term two (July 2024) will be obtained from the school to be used as pre-intervention and immediately post-intervention data for academic performance, respectively.
Height | Changes from baseline to immediately after the intervention and two month following the cessation of the intervention.
  Height will be measured in centimetres with a portable stadiometer.
Weight | Changes from baseline to immediately after the intervention and two month following the cessation of the intervention.
  Weight in kilograms will be determined with a Tanita device (Tanita Corp., Tokyo, Japan).
BMI | Changes from baseline to immediately after the intervention and two month following the cessation of the intervention.
  Weight and height will be combined to report BMI in kg/m^2
Waist circumference | Changes from baseline to immediately after the intervention and two month following the cessation of the intervention.
  Waist circumference in centimetres will be measured using a tape.
Body fat percentage | Changes from baseline to immediately after the intervention and two month following the cessation of the intervention.
  Body fat percentage will be determined with a Tanita device (Tanita Corp., Tokyo, Japan).
Physical activity | Baseline, first week and last week of the intervention and first week following the completion of the intervention.
  Physical activity for a subset of participants (n = 60) will be objectively assessed using GENEActiv wrist-worn accelerometers (Model GAT04, Activinsights Ltd, Cambridgeshire, England) over a span of four weeks, comprising one week before and after the intervention as well as the initial and concluding weeks of the intervention.
Bone health | Changes from baseline to immediately after the intervention and two month following the cessation of the intervention.
  A heel ultrasound test will be performed via a Achilles heel ultrasound machine (GE Medical Systems Lunar, USA). Participants will be seated with one foot on the foot plate, and alcohol will be applied to ensure proper membrane contact. A transducer on one side of the heel will convert an electrical signal into a sound wave, which will pass through the heel to the other side and be received and analysed by another transducer.
Perceived physical ability | Changes from baseline to immediately after the intervention and two month following the cessation of the intervention.
  A 6-item validated Perceived Physical Ability Scale will be utilised to evaluate the PA-related self-efficacy. The items are structured in response scales having a 1- to 4-point format. High scores would indicate a high self-perception of physical ability, whereas low scores would reflect a low self-perception.
Flanker task | Changes from baseline to immediately after the intervention and two month following the cessation of the intervention.
  Participants' inhibition will be assessed using a modified Flanker task. In the task, participants respond as quickly and accurately as possible to the direction of the fish in the middle which is flanked by another four fishes that are either swimming towards the same direction (congruent) or opposite direction (incongruent) to the central target fish. Participants will be instructed to press the "F" button on the keyboard if the fish swims towards left or "J" if towards right. The task consists of 104 trials in total, with a 1-minute rest when participants finished the first 52 trials. The result will be reported and compared as reaction time and accuracy.
Visual 2-back task | Changes from baseline to immediately after the intervention and two month following the cessation of the intervention.
  Working memory will be assessed using a modified visual 2-back task. Stimuli are sequences of animals (i.e., pig, giraffe, panda, snail and duck) which will be presented on the screen one-by-one. Participants will be instructed to respond to the stimulus as quickly and accurately as possible by either press the "F" button on the keyboard if the stimulus is identical to the one that appeared two trials back or "J" if not. The task consists of 52 trials in total, with a 1-minute rest when participants finished the first 26 trials. The result will be reported and compared as reaction time and accuracy.
Colour-shape switch task | Changes from baseline to immediately after the intervention and two month following the cessation of the intervention.
  Cognitive flexibility will be evaluated by a modified version of colour-shape switch task. In the task, participants will be instructed to react as quickly and accurately as possible to press the "F" button or "J" on the keyboard, with the following cues: If the object is at the top of the screen: press "F" if it is blue, press "J" if it is green; If the object is at the bottom of the screen: press "F" if it is square, press "J" if it is triangular. The task consists of 128 trials in total, with a 1-minute rest when participants finished the first 64 trials. The result will be reported and compared as reaction time and accuracy.

OTHER OUTCOMES:
Confounding variables | Maturity, subjectively measured physical activity and sleep will be measured at baseline, immediately after the intervention and two month following the cessation of the intervention.
  Age of peak height velocity will be used to assess the somatic maturation of participants. Participants' physical activity and sleep at all time-points will be assessed by a Chinese version of the International Physical Activity Questionnaire, short form and a validated Chinese version of the Pittsburgh Sleep Quality Index, respectively.
Interview | immediately after the intervention
  Semi-structured interviews will be conducted with participants and physical education teachers, separately, when the intervention completed. Pre-determined open questions will be asked during the interview, including feedback on enjoyment/usefulness of the intervention, continue performing/using the HIIT exercises and perceived barriers and facilitators for doing/delivering the HIIT exercises.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Williams, PhD, Study Chair — University of Exeter; Yaodong Gu, PhD, Study Chair — Ningbo University
Locations (1):
- University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu Y, Barker AR, Adlam AR, Li M, Duncombe SL, Agbaje AO, Gu Y, Zhou H, Williams CA. Effectiveness of a school-based high-intensity interval training intervention in adolescents: study protocol of the PRO-HIIT cluster randomised controlled trial. Front Pediatr. 2024 Oct 29;12:1458610. doi: 10.3389/fped.2024.1458610. eCollection 2024. PMID 39534248